CLINICAL TRIAL: NCT01239615
Title: Test-retest Stability of MR-parameters. A Neuroimaging Pilot-study in Healthy Volunteer
Brief Title: Test-retest Stability of MR-parameters. A Neuroimaging Pilot-study in Healthy Volunteers
Status: Withdrawn | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Søren Dinesen Østergaard, Associate Professor, Aarhus University Hospital
Other Study IDs: VEK-20100061
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Magnetic Resonance

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy volunteers

SUMMARY:
Aim: To study the stability of brain MR-scanning parameters (blood-flow, microstructure, volume, metabolism) over 1 week in health volunteers.

Hypothesis: MR-scanning parameters are stable over 1 week in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* oral and written consent

Exclusion Criteria:

* intracranial disease
* previous intracranial surgery
* magnetic implant or magnetic foreign body
* claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
cortical volume/thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg Hospital, Aalborg, Denmark